CLINICAL TRIAL: NCT01236703
Title: Hematological Infection Profile (ICIS/ICPS) Compared to Actual Best Hospital Practice for Differentiation of SIRS and Sepsis and Management of Antiinfective Therapy in ICU Patients
Brief Title: Hematological Infection Score Compared to the Hospital Standard for Diagnosis of SIRS or Sepsis on ICU
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Sysmex Europe GmbH (Industry)
Responsible Party: Principal Investigator, Claudia Spies, Univ. Prof. Dr. med. Claudia Spies, Charite University, Berlin, Germany
Other Study IDs: HemoSIRS
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: SIRS; Sepsis
Keywords: SIRS; Sepsis; hematological infection score
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: ICU patients (post-operative and none operative patients) will be enrolled in the study. They are followed up until the end of ICU stay or, for a maximum of 60 days.

SUMMARY:
CRP and PCT are not valid parameters of early infection in particularly postoperative patients. (Sanders et al., A&A, June 2006, Vol.102; Katja et al., Shock, February 2001, Vol 15.2) Better detection systems for SIRS and sepsis are urgently required.

ICIS® (Sysmex intensive care infection score) and ICPS® (Sysmex intensive care prognostic score) are two new score-systems depending on detectable cellular response of the innate immune system in human peripheral blood.

The purpose of this observational study is to determine if these scores are superior in early differentiation between non-infectious SIRS and infectious SIRS (sepsis) in postoperative patients. Furthermore, the applicability of the scores for triggering start and ending of anti-infective therapy will be examined.

ELIGIBILITY:
Inclusion Criteria:

* all ICU patients age > 18 years
* more than 36h on ICU

Exclusion Criteria:

* ICU patients age < 18 years
* less than 36h on ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All IC department patients (WAN 8i, WAN 14i and WNC S1i Charite Berlin) will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study performed according to an observational post-ad-hoc design is to show that the two Sysmex infection scores provide a better performance than CRP & PCT for infection processes thus providing an efficient alternative. | a period of 60 days
  Approximately 200 patients will be enrolled in the study. They are followed up until the end of ICU stay or, for a maximum of 60 days. Usually in clinical routine, patients suspected to have an infection process, receive once per day a "full infectiology profile". It consists of CRP, PCT and the Sysmex infection profiles (ICIS/ICPS).

SECONDARY OUTCOMES:
The second objective is to investigate whether ICIS® and ICPS® could assist in faster antiinfective regim decisions than CRP & PCT. | a period of 60 day
  Approximately 200 patients will be enrolled in the study. They are followed up until the end of ICU stay or, for a maximum of 60 days. Usually in clinical routine, patients suspected to have an infection process, receive once per day a "full infectiology profile". It consists of CRP, PCT and the Sysmex infection profiles (ICIS/ICPS).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Department of Anesthesiology and Operative Intensive Care Medicine Campus Virchow-Klinikum, Berlin, State of Berlin, Germany